CLINICAL TRIAL: NCT00475046
Title: Smoking Cessation and Relapse Prevention in Women Postpartum
Acronym: EARLINT-EP3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01EB0120-TP3
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Smoking Cessation
Keywords: smoking; post partum; relapse prevention; motivational interviewing; TTM; implement motivational enhancement interventions in pediatric practices; examine the effectiveness of the intervention; develop measurements appropriate to tailor interventions; analyze further unfavorable and favorable factors outlined by previous research
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Motivational Interviewing

SUMMARY:
Background: Pregnancy was found to be a significant triggering factor for smoking cessation and the reduction of nicotine consumption, but 50 - 70 % of mothers who stopped smoking during pregnancy resume tobacco smoking after delivery. One main reason for the high relapse rates is that many women are solely motivated to quit smoking for the baby's sake. After birth, the external reason for having quit has vanished and no other internal or external motives exist for many women to maintain being smoke-free. Therefore, under consideration of the Transtheoretical Model approach, relapse prevention and smoking cessation interventions have to focus on two aspects: (1) on a specific reformulation of the stages of change for women who show a temporarily and externally motivated change in smoking behavior during pregnancy, (2) on intervention strategies taking advantage of the behavioral change already done and evoking the cognitive and behavioral processes necessary for maintenance. In Germany pediatricians are in a unique position to address this issue because nearly every mother attends a pediatric practice for preventive examination of the newborn. Objectives: To adapt and implement motivational enhancement interventions in pediatric practices. The aim is to examine the effectiveness of a modified stage-matched motivational enhancement intervention added to the common pediatricians´ advice. A second aim is the reformulation and reassessment of the stages of change for women who have recently given birth. Methods: The study design is a randomized controlled trial. Mothers smoking at the beginning of the pregnancy and attending pediatric practices in West Pomerania will be assigned to an intervention group (n = 330) and referred to a liaisonal service providing a face-to-face motivational enhancement intervention followed by telephone brush-up sessions. A control group (n = 330) receives treatment from the pediatrician as usual at the preventive examination. The core outcome measures comprise abstinence, and progress in the stages of change 6, 12, 18 and 24 months after baseline. Expected impact: Data will evaluate the usefulness of intervening in pediatric offices and will provide information about a tailored intervention program. The processes of change favorable for intervention in this population will be identified. This is of great relevance with regard to the prevention of health damage for mother and child. Furthermore, results will serve as a basis for guidelines for pediatricians to deal with women smoking postpartum. Relationship to the objective of the collaboration: As in the other studies, this study provides empirical data of a new proactive approach to reach underserved populations in the addiction field. This project will add knowledge on how to intervene (motivational enhancement vs. usual advice), on setting-specific advantages of pediatric offices and on the impact of the chosen intervention strategy.

DETAILED DESCRIPTION:
5.1.1 Sample The 526,761-inhabitant region of West Pomerania comprises 28 pediatric practices. Every mother presenting her newborn for the first time in the pediatric practices will be screened. Of these, all women smoking at the date the female received verification of her pregnancy are eligible for the study. A power analysis on grounds of data from Johnson et al. (2000) and using the software nquery (Elashoff, 2000) revealed that a sample size of 259 women per group will provide a power of 80 % using the five percent one-tailed significance level to compare the experimental and the control group with regard to the prevalence of sustained smoking abstinence 6 months after intervention by a two groups continuity corrected Chi2-test of equal proportions. Assuming an attrition of approximately 25 %, it results in a sample size of 330 women per group. According to the statistical regional authorities of the mentioned region, 3,527 babies were born alive in the year 1998. Therefore 1,234 mothers smoking at the beginning of pregnancy (35 %) per year are expected. Assuming a pediatric practice participation rate of 70 % and an 80 % participation rate of women eligible for the study, about one year of data gathering will be necessary to reach the estimated total sample size of 660 mothers.

5.1.2 Procedure Procedure of the study This study is a randomized controlled trial following a repeated measures factorial design and enabling the comparison of one intervention group with a control group. The work plan of the study incorporates 6 months of preparatory work including the adaptation of instruments for the assessment of core constructs of the Transtheoretical Model and a pre-test, 12 months of screening by receptionists in pediatric practice and the recruitment of eligible women for the study by the pediatrician after giving written informed consent (figure 1). Random assignment to control and intervention group will be done after forwarding the women's addresses to the liaisonal service provided by research staff. The intervention phase of the study will be completed 6 months after the last recruitment. Follow-ups will be carried out 6, 12, 18 and 24 months after baseline assessment. Data analyses and publication will be started in the third year. Analysis of the 18 and 24 month data will exceed the three year period of support.

Figure 1: Time schedule postpartum tobacco smoking relapse prevention intervention

Procedure for participants Figure 2 details the succession of steps for participants. Every woman at her first postpartum visit to a pediatric practice (usually 4 to 6 weeks after giving birth) will be screened by receptionists concerning her smoking status, considering the time at the beginning of the pregnancy, and informed about the study by the pediatrician. All participants will receive treatment as usual at the time of preventive examination of newborns by the pediatrician. After baseline assessment by phone, the intervention group will receive an initial face-to-face counseling at home one week after the pediatric practice visit at home. Two brush-up counseling sessions will be provided by phone 3 and 6 months later. Follow-up assessment will be conducted by phone.

Figure 2: Procedure for participants

5.1.3 Intervention In the intervention group, motivational interviewing will be conducted by psychologists qualified by a comprehensive training curriculum offered at the University of Greifswald according to Miller & Rollnick (1991). Face-to-face and phone counseling will be tailored by data from baseline assessment and are conceived for a duration of up to 45 minutes. A tailored information and self-help manual will be given at the initial counseling. If the allowance of the participant is received, a tape recording of a random selection of counseling sessions will be done for intervention control. The control group will receive advice as usual from the pediatrician.

5.1.4 Measures To ensure cross-study comparison, all measures will be operationalized by internationally standardized and validated state of the art instruments, if available.

Pre-intervention measures

* pregnancy history
* smoking behavior and history, severity of nicotine dependence
* environmental smoking
* health behavior
* child health
* Adapted Transtheoretical Model core constructs (Stage allocation, processes of change, decisional balance, and temptation/self-efficacy) based on previous work of Ruggiero et al. (2000) and Bane et al. (1999).

Post-intervention measure

* Current and sustained smoking abstinence prevalence, amount of cigarettes smoked per day
* Adapted Transtheoretical Model core constructs

Statistical analysis for the main outcome measure will be done by Chi²-test, T-test and repeated measure MANOVA. Outcome predictors will be analyzed by logistic regression analysis.

5.2 Collaboration 5.2.1 Within EARLINT There will be a close cooperation within EARLINT with all studies comprising motivational enhancement intervention by personal counseling. Quality assurance and training curricula will be matched for all projects.

5.2.2 External This study will be conducted in cooperation with pediatric offices in West Pomerania. Contact has been established with the regional professional organization of pediatricians and Prof. Fusch (Department for Pediatrics at the University of Greifswald). Further collaboration exists with the only research group with comparable work in Germany (Dr. Lang, Prof. Greiser, University of Bremen).

5.3 Ethical and legal correctness All ethical and legal safeguards have been met. The study is currently being refereed by the local ethical committee. The study involves no risk to participants. To the contrary, health benefits are expected. Individuals will be informed of their right to refuse to participate in any or all aspects of the study and will be given opportunities to terminate enrollment. Informed consent forms and an introductory letter will assure individuals that their participation is voluntary and that data protection laws have been met.

ELIGIBILITY:
Inclusion Criteria:

* Every mother presenting her newborn for the first time in the pediatric practices will be screened. Of these, all women smoking at the date the female received verification of her pregnancy are eligible for the study.

Min Age: 1 Year | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2790 (Actual)
Dates: Start 2001-10; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Current and sustained smoking abstinence prevalence, amount of cigarettes smoked per day | 6, 12, 18 and 24 monthy after baseline

SECONDARY OUTCOMES:
Adapted Transtheoretical Model core constructs | 6, 12, 18 and 24 monthy after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ulfert Hapke, PhD, Principal Investigator — Institut für Epidemiologie und Sozialmedizin, University of Greifswald

REFERENCES:
- [Background] Hannover W, Thyrian JR, Roske K, Kelbsch J, John U, Hapke U. [Interventions to prevent health risks due to tobacco smoke in pregnant women, postpartum women and their infants]. Gesundheitswesen. 2004 Oct;66(10):688-96. doi: 10.1055/s-2004-813602. German. PMID 15499514
- [Background] Hannover W, Thyrian JR, John U. Short report: Paediatricians' attitude towards counselling parents postpartum about their smoking behaviour. Eur J Public Health. 2004 Jun;14(2):199-200. doi: 10.1093/eurpub/14.2.199. PMID 15230510
- [Background] Roske K, Hannover W, Kelbsch J, Thyrian JR, John U, Hapke U. [The readiness of women, after they have given birth to children, to participate in individualized counselling for smoking cessation ]. Gesundheitswesen. 2004 Oct;66(10):697-702. doi: 10.1055/s-2004-813621. German. PMID 15499515
- [Background] Thyrian JR, Hanke M, Hannover W, Grempler J, Roske K, Fusch C, John U. [Exposure to tobacco smoke (passive smoking) in the home and inpatient treatment of children under the age of 5 years in Germany]. Dtsch Med Wochenschr. 2005 May 13;130(19):1189-94. doi: 10.1055/s-2005-868699. German. PMID 15875260
- [Background] Roske K, Hannover W, Grempler J, Thyrian JR, Rumpf HJ, John U, Hapke U. Post-partum intention to resume smoking. Health Educ Res. 2006 Jun;21(3):386-92. doi: 10.1093/her/cyh069. Epub 2005 Nov 17. PMID 16293673
- [Background] Thyrian JR, Hannover W, Grempler J, Roske K, John U, Hapke U. An intervention to support postpartum women to quit smoking or remain smoke-free. J Midwifery Womens Health. 2006 Jan-Feb;51(1):45-50. doi: 10.1016/j.jmwh.2005.07.002. PMID 16399610
- [Background] Thyrian JR, Hannover W, Roske K, Rumpf HJ, John U, Hapke U. Postpartum return to smoking: identifying different groups to tailor interventions. Addict Behav. 2006 Oct;31(10):1785-96. doi: 10.1016/j.addbeh.2005.12.016. Epub 2006 Jan 23. PMID 16431031
- [Background] Thyrian JR, Hannover W, Roske K, Scherbarth S, Hapke U, John U. Midwives' attitudes to counselling women about their smoking behaviour during pregnancy and postpartum. Midwifery. 2006 Mar;22(1):32-9. doi: 10.1016/j.midw.2005.04.003. PMID 16488809
- [Background] Roske K, Hannover W, Thyrian JR, Grempler J, Rumpf HJ, John U, Hapke U. [Why woman postpartum resume smoking]. Gesundheitswesen. 2006 Mar;68(3):171-5. doi: 10.1055/s-2006-926639. German. PMID 16575697
- [Background] John U, Meyer C, Ulbricht S, Schumann A, Freyer-Adam J, Hapke U, Rumpf HJ, Bischof G, Grothues J, Thyrian JR. [Improvement of medical care by supporting the intention to change health risk behavior]. Med Klin (Munich). 2007 Jan 15;102(1):33-6. doi: 10.1007/s00063-007-1006-7. German. PMID 17221350
- [Background] Thyrian JR, Freyer-Adam J, Hannover W, Roske K, Mentzel F, Kufeld C, Bischof G, Rumpf HJ, John U, Hapke U. Adherence to the principles of Motivational Interviewing, clients' characteristics and behavior outcome in a smoking cessation and relapse prevention trial in women postpartum. Addict Behav. 2007 Oct;32(10):2297-303. doi: 10.1016/j.addbeh.2007.01.024. Epub 2007 Jan 23. PMID 17307300
- [Background] Thyrian JR, Hannover W, Roske K, John U, Hapke U. Smoking before, during and after pregnancy: Longitudinal data from a population-based sample. Geburtshilfe Und Frauenheilkunde, 65(7), 687-689